CLINICAL TRIAL: NCT00000782
Title: A Phase I/II Study of Delayed-Type Hypersensitivity (DTH) Reactions to Intradermal HIV Envelope Antigen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 221; 11198 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Injections, Intradermal; HIV Antigens; HIV-1; HIV Envelope Protein gp160; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Hypersensitivity, Delayed; AIDS Vaccines; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Hypersensitivity, Delayed | interventions — VaxSyn HIV-1 (gp160) vaccine

INTERVENTIONS:
Biological: gp160 Vaccine (Immuno-AG)
Biological: gp160 Vaccine (MicroGeneSys)

SUMMARY:
To determine the frequency of delayed-type hypersensitivity (DTH) reactions in HIV-positive patients to two doses of two envelope glycoprotein antigens prepared differently. To determine whether patients who have previously demonstrated a DTH response to intradermal MGStage HIV-1 gp160 IIIB baculovirus (MicroGeneSys) have a reproducible response to a repeat injection of gp160 and whether there is cross-reactivity to intradermal HIV-1 rgp160 IIIB vero cell expressed (Immuno-AG).

PER 4/5/95 AMENDMENT: To also determine whether patients who respond to HIV-1 rgp160 IIIB baculovirus (MicroGeneSys) have cross-reactivity to intradermal skin tests of HIV-1 rgp160 MN (Immuno-AG).

Previous studies in individuals immunized with gp160 suggest that a skin test response in immunized patients can be used as a surrogate marker for new proliferative and cytotoxic responses induced by vaccination.

DETAILED DESCRIPTION:
Previous studies in individuals immunized with gp160 suggest that a skin test response in immunized patients can be used as a surrogate marker for new proliferative and cytotoxic responses induced by vaccination.

Patients are stratified into three groups. Fifteen patients previously immunized with MicroGeneSys rgp160 antigen in ACTG 137 and not on antiretroviral therapy will receive intradermal injections of Immuno-AG rgp160 IIIB (vero cell expressed) in one arm, followed 1 week later by intradermal injections of MicroGeneSys rgp160 IIIB (baculovirus expressed) in the opposite arm (stratum 1). Forty patients who are not previously immunized with rgp160 will receive intradermal injections of Immuno-AG gp160 IIIB in one arm simultaneously with MicroGeneSys gp160 IIIB in the opposite arm; these patients are either not on antiretroviral therapy (stratum 2) or currently on antiretroviral therapy (stratum 3). All patients return 48 hours after each injection for skin test reading.

PER 4/5/95 AMENDMENT: Patients on all strata will re-enroll to receive Immuno-AG rgp160 MN in one arm simultaneously with MicroGeneSys rgp160 IIIB in the opposite arm.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed in Step 2 (PER 4/5/95 AMENDMENT):

* Approved antiretroviral drugs.

Patients must have:

* Documented HIV infection.
* CD4 count >= 400 cells/mm3.
* NO current active opportunistic infection or neoplasm (other than stable cutaneous Kaposi's sarcoma).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known hypersensitivity to insect proteins.

Concurrent Medication:

Excluded:

* Antihistamine or anti-inflammatory medications for the 48-hour period between injection and skin test reading.
* Topical steroids.

Prior Medication:

PER 4/5/95 AMENDMENT -

Excluded:

* Prior immunization with experimental HIV vaccines (strata 2 and 3 only).
* Systemic corticosteroids, topical corticosteroids on the arms, or other systemic immunosuppressant agents or antineoplastic agents within 30 days prior to study entry.
* Antihistamine or anti-inflammatory medications within 72 hours prior to intradermal injections.

PREVIOUS VERSION -

Excluded within 30 days prior to study entry:

* Any antiretroviral drugs (other than AZT, ddI, ddC, or d4T for patients in stratum 3).
* Systemic corticosteroids, topical corticosteroids on the arms, or other systemic immunosuppressant agents or antineoplastic agents.

Excluded within 72 hours prior to intradermal injections:

* Antihistamine or anti-inflammatory medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Study Completion 1996-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katzenstein D, Study Chair
Locations (4):
- United States (4):
  - Stanford CRS, Palo Alto, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - NY Univ. HIV/AIDS CRS, New York, New York

REFERENCES:
- [Background] Katzenstein DA, Kundu S, Spritzler J, Smoller BR, Haszlett P, Valentine F, Merigan TC. Delayed-type hypersensitivity to recombinant HIV envelope glycoprotein (rgp160) after immunization with homologous antigen. J Acquir Immune Defic Syndr. 1999 Dec 1;22(4):341-7. doi: 10.1097/00126334-199912010-00004. PMID 10634195